CLINICAL TRIAL: NCT01222260
Title: Phase II Study of the Combination of Bendamustine and Dexamethasone in Patients With Relapsed AL Amyloidosis
Brief Title: Bendamustine and Dexamethasone in Patients With Relapsed AL Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Principal Investigator, Suzanne Lentzsch, MD, Associate Professor of Clinical Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAJ7800; 10-012 (PRO10050217) (Other: University of Pittsburgh)
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Results first posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: AL Amyloidosis
Keywords: Amyloidosis; Dexamethasone; Bendamustine; Relapsed AL Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Amyloidosis | interventions — Bendamustine Hydrochloride; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Arm (Experimental): Subjects with AL will receive Bendamustine and Dexamethasone
  Interventions: Drug: Bendamustine; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bendamustine — Patients will start bendamustine at dose level 0 and according to CrCl on day 1 and 2 of each cycle:
  * CrCl ≥ 60 mL/min: 100 mg/m2 IV on day 1 and 2 of each cycle
  * CrCl 59 - 30 mL/min: 90 mg/m2 IV on day 1 and 2 of each cycle
  Available to qualifying subjects is the option to dose escalate to dose level (+)1:
  * 120 mg/m2 (if CrCl ≥ 60 mL/min at the time of inclusion into the study)
  * 100 mg/m2 (if CrCl 59-30 mL/min at the time of inclusion into the study)
  Other Names: Bendamustine Hydrochloride; Treanda ®
Drug: Dexamethasone — 40 mg orally on days 1, 8, 15, 22 of each cycle
  Other Names: Decadron

SUMMARY:
The study is being done to see if the combination of bendamustine and dexamethasone will help people with amyloidosis that has returned after standard treatment, and to to estimate the partial hematologic response rate (PHR).

DETAILED DESCRIPTION:
Systemic light-chain amyloidosis (AL) is a protein conformation disorder due to a clonal plasma cell dyscrasia. There are no established and approved second-line therapies for patients with systemic AL amyloidosis who fail initial melphalan-based treatment, be it high-dose melphalan with stem cell transplant or oral melphalan and dexamethasone (MDex). Therefore new treatments are needed for those who fail initial therapy and for those who initially respond but subsequently relapse.

Therapy of AL is generally based on treatment regimens used in multiple myeloma (MM). Bendamustine achieves partial response with relapsed/refractory MM. Based on this high anti-MM activity, we anticipate that bendamustine will also be very active in clonal plasma cell disorder associated with AL.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 18 years old
* Histopathology of amyloidosis or light chain deposition disease based on detection by polarizing microscopy of green bi-refringent material in Congo red-stained tissue specimens or characteristic electron microscopy appearance or immunohistochemical stain with anti-light chain anti-sera
* Demonstrate measurable disease as defined by one or more of the following:

  * Serum monoclonal protein ≥ 0.5 g/dL by serum electrophoresis
  * Urine monoclonal protein > 200 mg/dL in a 24 hr urine electrophoresis
  * Serum immunoglobulin free light chain ≥ 5 mg/dL and abnormal serum immunoglobulin kappa lambda free light chain ratio. The difference between involved and uninvolved free light chains should be ≥ 5 mg/dL (dFLC)
  * Demonstrate clonal population of plasma cells in the bone marrow or immunohistochemical stain with anti-light chain anti-sera of amyloid fibrils
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Patients had at least one prior regimen consisting of at least 1 cycle
* If not previously transplanted, patient should be either ineligible for autologous stem cell transplantation (ASCT), or must have declined the option of ASCT. Patients who have previously had ASCT and have subsequently progressed are eligible, provided other entry criteria are met
* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed

Patients must meet the following laboratory criteria:

* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
* Hemoglobin ≥ 9 g/dl (May transfuse packed red blood cells (PRBC) to meet parameter)
* Platelets ≥ 100x 10^9/L (Must be independent of platelet transfusion)
* Calculated creatinine clearance (CrCl) greater than or equal to 30 mL/min (Cockcroft-Gault Formula )
* Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x upper limit of normal (ULN)
* Serum bilirubin <1.5 x ULN
* Serum potassium within normal limits
* Total serum calcium (corrected for serum albumin) or ionized calcium ≤ ULN

Exclusion Criteria:

* Patients meeting the criteria for symptomatic MM:
* Lytic lesions on skeletal survey or plasmacytoma

Patients meeting International Myeloma Working Group definition of symptomatic myeloma with symptoms only related to associated amyloidosis who would otherwise only meet the criteria for smoldering MM are potentially eligible

* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure uncontrolled angina, severe uncontrolled ventricular arrhythmias, or
* electrocardiographic evidence of acute ischemia or active conduction system abnormalities (not including 1st degree atrioventricular (AV)-block, Wenckebach type 2nd degree heart block, or left bundle branch block. Prior to study entry, any electrocardiogram (ECG) abnormality at Screening has to be documented by the investigator or an authorized physician sub-investigator as not medically relevant). Note: There is no lower limit of left ventricular ejection fraction below which patients are excluded from participation.
* Patients with N-terminal (NT)-proBNP ≥ 1800nb/L or B-type natriuretic peptide (BNP) ≥ 400 ng/L, abnormal cardiac troponin T (cTnT) or cardiac troponin l (cTnI)
* Patient has received other investigational drugs within 14 days prior to enrollment
* Any form of secondary / familial amyloidosis
* Serious concurrent illness, which in the opinion of the investigator or an authorized physician sub-investigator would interfere with participation in this clinical study,
* Known HIV infection.
* Inability to provide informed consent or to comply with the schedule of office and treatment visits
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women(woman not of child-bearing potential is defined as any woman whose menstrual periods have stopped in the past 12 consecutive months or have had a complete hysterectomy or both ovaries surgically removed).
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, low-risk prostate cancer, or cancer after curative treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Lentzsch, MD, PhD, Principal Investigator — Columbia University
Locations (6):
- United States (6):
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mt. Sinai Medical Center, New York, New York
  - Columbia University, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data that underlie the reported results will be made available 3 months after publication for a period of 5 years after the publication.
Supporting Information: Study Protocol
Time Frame: 3 months after manuscript publication for a period of 5 years after the publication.
Access Criteria: Proposals for access should be sent to cancerclinicaltrials@cumc.columbia.edu.

REFERENCES:
- [Derived] Lentzsch S, Lagos GG, Comenzo RL, Zonder JA, Osman K, Pan S, Bhutani D, Pregja S, Sanchorawala V, Landau H. Bendamustine With Dexamethasone in Relapsed/Refractory Systemic Light-Chain Amyloidosis: Results of a Phase II Study. J Clin Oncol. 2020 May 1;38(13):1455-1462. doi: 10.1200/JCO.19.01721. Epub 2020 Feb 21. PMID 32083996

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between January 2013 and March 2016, 40 patients were enrolled in the study and 31 patients were treated.
Groups:
- Treatment Arm: Subjects with relapsed/refractory systemic light-chain (AL) will receive Bendamustine and Dexamethasone.
  Bendamustine: Patients will start bendamustine at dose level 0 and according to creatinine clearance (CrCl) on day 1 and 2 of each cycle:
  * CrCl ≥ 60 mL/min: 100 mg/m2 IV on day 1 and 2 of each cycle
  * CrCl 59 - 30 mL/min: 90 mg/m2 IV on day 1 and 2 of each cycle
  Available to qualifying subjects is the option to dose escalate to dose level (+)1:
  * 120 mg/m2 (if CrCl ≥ 60 mL/min at the time of inclusion into the study)
  * 100 mg/m2 (if CrCl 59-30 mL/min at the time of inclusion into the study)
  Dexamethasone: 40 mg orally on days 1, 8, 15, 22 of each cycle
Period: Overall Study
Arm/Group | Treatment Arm
Started | 31
Completed | 29
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm: Subjects with AL will receive Bendamustine and Dexamethasone
  Bendamustine: Patients will start bendamustine at dose level 0 and according to CrCl on day 1 and 2 of each cycle:
  * CrCl ≥ 60 mL/min: 100 mg/m2 IV on day 1 and 2 of each cycle
  * CrCl 59 - 30 mL/min: 90 mg/m2 IV on day 1 and 2 of each cycle
  Available to qualifying subjects is the option to dose escalate to dose level (+)1:
  * 120 mg/m2 (if CrCl ≥ 60 mL/min at the time of inclusion into the study)
  * 100 mg/m2 (if CrCl 59-30 mL/min at the time of inclusion into the study)
  Dexamethasone: 40 mg orally on days 1, 8, 15, 22 of each cycle
Arm/Group | Treatment Arm
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: years] | 65 [42 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 15
  More than one race | 0
  Unknown or Not Reported | 13
Time since diagnosis [Median (Full Range); unit: months] | 31.0 [3.0 to 167.2]

OUTCOME MEASURES:

1. Primary Outcome: Partial Hematologic Response (PHR) Rate
Description: Only patients who have received at least 2 cycles of therapy are eligible for response assessment. The proportion of patients with PHR two months post-treatment will be estimated, with a 95% exact binomial confidence interval. Partial response is defined as the reduction of the difference between involved and uninvolved free light chains (dFLC) of ≥ 50% OR a reduction of ≥ 50% of the M-protein if M-spike is ≥ 0.5 g/dL.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 28
Participants | 16

2. Secondary Outcome: Overall Hematologic Response Rate (OHR)
Description: The proportion of response-evaluable patients experiencing OHR will be estimated, with a 95% exact binomial confidence interval. Overall hematologic response rate as defined by normalization of the free light chain levels and ratio, negative serum and urine immunofixation OR reduction in the difference between involved and uninvolved free light chains (dFLC) to <4 mg/dL.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 28
Participants | 16

3. Secondary Outcome: Organ Response Rate (ORR)
Description: The proportion of response-evaluable patients experiencing ORR will be estimated, with a 95% exact binomial confidence interval. Amyloid-related organ response will be evaluated on the basis of the accepted criteria described: Kidneys: 30% reduction or drop below 0.5 g in 24-hour urine protein excretion in the absence of progressive renal insufficiency. Heart: N-terminal pro b-type natriuretic peptide (NT-proBNP) or B-type natriuretic peptide response (>30% and >300 ng/L decrease in patients with baseline NT-proBNP ≥ 650 ng/L or New York Heart Association (NYHA) class response (≥ 2 class decrease in subjects with baseline NYHA class 3 or 4). Liver: 50% decrease of an initially elevated alkaline phosphatase level or reduction in the size of the liver by at least 2 cm. Neuropathy: improvement supported by clinical history, neurologic exam, orthostatic vital signs, resolution of severe constipation or reduction of diarrhea to less than 50% of previous movements/day.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 24
Participants | 7

4. Secondary Outcome: Median Overall Survival (OS)
Description: Survival is assessed as time to death from first day of treatment The OS function for response-evaluable will be estimated using the product-limit (Kaplan-Meier) estimator, along with 95% confidence bounds. The median survival will be estimated from the survival function. The analysis will be repeated on all patients who receive any therapy.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment Arm
Number analyzed (Participants) | 28
months | 18.2 [11.3 to 43.8]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 1/29
Serious Adverse Events (participants affected / at risk) | 10/29
Other Adverse Events (participants affected / at risk) | 20/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=29)
Fatigue (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Renal dysfunction (Renal and urinary disorders) | 2 (2)
Infection (Infections and infestations) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Infusion-related reaction (General disorders) | 1 (1)
Fever and chills (Infections and infestations) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=29)
Fatigue (General disorders) | 8 (8) — Grade 3
Decreased lymphocyte count (Blood and lymphatic system disorders) | 6 (6) — Grade 3
Chronic kidney disease (Renal and urinary disorders) | 4 (4) — Grade 3
Hypotension (General disorders) | 3 (3) — Grade 3
Hypertension (General disorders) | 3 (3) — Grade 3
Decreased neutrophil count (Blood and lymphatic system disorders) | 3 (3) — Grade 3
Syncope (General disorders) | 3 (3) — Grade 3
Nausea (General disorders) | 2 (2) — Grade 3
Decreased white blood cell count (Blood and lymphatic system disorders) | 2 (2) — Grade 3
Anemia (Blood and lymphatic system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-03): https://cdn.clinicaltrials.gov/large-docs/60/NCT01222260/Prot_SAP_000.pdf